CLINICAL TRIAL: NCT00074009
Title: A Multicenter, Open-Label, Two-Stage, Phase II Study Of PS-341 (LDP-341, NSC # 681239) In Patients With Unresectable Or Metastatic Gastric Adenocarcinoma
Brief Title: Bortezomib in Treating Patients With Unresectable or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000341565; MSKCC-03101; NCI-6003
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2009-12

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have unresectable or metastatic gastric cancer or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of bortezomib in patients with unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.

Secondary

* Determine the toxicity of this drug in these patients.
* Determine possible predictors of response to this drug, using pretreatment tumor immunohistochemistry, in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 15-33 patients will be accrued for this study within 5-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma

  * Siewert's class II or III disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No history of known or active brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100% OR
* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No prior cerebrovascular event
* No prior orthostatic hypotension
* No myocardial infarction within the past 6 months
* No peripheral vascular disease requiring surgical management
* No evidence of acute ischemia or significant conduction abnormality by EKG

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after study participation
* No evidence of peripheral neuropathy
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to bortezomib
* No other malignancy within the past 3 years except basal cell skin cancer, carcinoma in situ of the cervix, or adequately treated nonmetastatic prostate cancer
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other concurrent uncontrolled illness that would preclude study participation
* No other medical condition or reason that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 weeks since prior immunotherapy
* No concurrent biological or immunological agents

Chemotherapy

* No more than 1 prior chemotherapy regimen (including adjuvant chemotherapy)
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* Recovered from all prior therapy
* No other concurrent investigational agents
* No other concurrent anticancer agent or therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish A. Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Gary K. Schwartz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Shah MA, Power DG, Kindler HL, Holen KD, Kemeny MM, Ilson DH, Tang L, Capanu M, Wright JJ, Kelsen DP. A multicenter, phase II study of bortezomib (PS-341) in patients with unresectable or metastatic gastric and gastroesophageal junction adenocarcinoma. Invest New Drugs. 2011 Dec;29(6):1475-81. doi: 10.1007/s10637-010-9474-7. Epub 2010 Jun 25. PMID 20574790